CLINICAL TRIAL: NCT05188963
Title: A Randomized Control Trial About Two Different Regimens of Clean Intermittent Catheterization in Women With Overt PUR: the DICOPUR Trial
Brief Title: RCT About Two Different Regimens of Clean Intermittent Catheterization in Women With Overt Postpartum Urinary Retention
Acronym: DICOPUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Soren Lange, Fellow, Principal Investigator, M.D., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1093/2021
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Urinary Retention; Postpartum Period
Keywords: postpartum urinary retention; intermittent catheterization; postvoid residual volume; postpartum
MeSH Terms: conditions — Urinary Retention | interventions — Intermittent Urethral Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women with postvoid residual volume cut-off at 150 ml (Active Comparator)
  Interventions: Procedure: Intermittent catheterization
- Women with postvoid residual volume cut-off at 250 ml (Experimental)
  Interventions: Procedure: Intermittent catheterization

INTERVENTIONS:
Procedure: Intermittent catheterization — Intermittent catheterization is performed as treatment for urinary retention. Treatment is stopped when postvoid urinary retention volume is below the threshold of each group.

SUMMARY:
A randomized controlled trial of two different regimens of intermittent catheterization in women with overt postpartum urinary retention.

Participants will be randomized to one of two groups with different cut-offs for accepted postvoid residual urine (150 ml vs 250 ml).

Primary endpoint is be the time to regain normal bladder function in each group. Secondary endpoints are 1) presence/absence of bacteriuria or urinary tract infections, 2) the duration of hospital stay, 3) scores on the adapted version of the German pelvic floor questionnaire section about bladder function and postpartum symptoms.

The calculated sample size is 96 (48 in each group).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed overt postpartum urinary retention.
* Age ≥ 18 years at delivery date.
* Delivery at study site.
* signed informed consent.

Exclusion Criteria:

* Refusal to participate.
* Language barrier.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Time to regain normal bladder function | 3 months
  The time until bladder function returned to normal.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna/Allgemeines Krankenhaus Wien, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No